CLINICAL TRIAL: NCT00389948
Title: A Phase III, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Trial of 14 Day Treatment With Lansoprazole 15 mg Once a Day in Frequent Heartburn
Brief Title: Efficacy/Safety of Lansoprazole in Patients With Frequent Heartburn
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRSW-GN-301
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2007-04-16 (Estimated); Status verified 2007-04

CONDITIONS: Heartburn
Keywords: Heartburn, frequent heartburn, proton pump inhibitor, lansoprazole
MeSH Terms: conditions — Heartburn

INTERVENTIONS:
Drug: Lanzoprazole

SUMMARY:
Heartburn, a burning sensation in the chest or throat, occurs in many patients when acidic stomach contents move into the esophagus from the stomach. This study will investigate the safety and efficacy of lansoprazole 15 mg once a day in treating frequent heartburn.

ELIGIBILITY:
Inclusion Criteria:

1. Experiencing heartburn at least 2 days per week over the past month.
2. Having heartburn that responds to heartburn medication.
3. Be willing to discontinue the use of heartburn treatment for 7 days prior to inclusion in the study.

Exclusion Criteria:

1. Having history of erosive esophagitis or gastroesophageal reflux disease diagnosed by a physician and confirmed by testing (endoscopy).
2. Be unwilling to take only the study medication, and antacid provided as a rescue medication for relief of acute heartburn during the study.

Other protocol-defined inclusion or exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576
Dates: Start 2006-06; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
To demonstrate that repeated daily doses of 15 mg of lansoprazole are effective in increasing the proportion of days with no heartburn during study treatment, when compared to placebo.

SECONDARY OUTCOMES:
To determine the proportion of nighttimes with no heartburn during 14 days of treatment in subjects receiving lansoprazole versus placebo
To determine the proportion of subjects with no heartburn during day 1 in those receiving lansoprazole versus placebo
Evaluation of lansoprazole safety.

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Clinical Research Consultants Inc., Hoover, Alabama
  - Huntsville, Alabama
  - Radiant Research, Sierra Vista, Arizona
  - California Bio Medical Research Institute, Los Angeles, California
  - Allergy Medical Group of North Area, Roseville, California
  - Eastern Research, Hialeah, Florida
  - Health Awareness Inc., Jupiter, Florida
  - Miami Research Associates, Miami, Florida
  - Radiant Research, Atlanta, Georgia
  - Evansville, Indiana
  - Clinical Associates, Reisterstown, Maryland
  - Medex Healthcare Research, Inc., St Louis, Missouri
  - Meridian Clinical Research LLC, Omaha, Nebraska
  - William W. Anderson M.D. P.C., Rio Rancho, New Mexico
  - IRSI, Port Chester, New York
  - Crescent Medical Research, Salisbury, North Carolina
  - Micheal Alexander, DO, Columbus, Ohio
  - New Hope Research of Oregon, Portland, Oregon
  - Preferred Primary Care Physicians, Carnegie, Pennsylvania
  - Advanced Therapeutics, Inc, Johnson City, Tennessee
  - Nashville Medical Research, Nashville, Tennessee
  - Medical Edge Healthcare Group, P.A., Dallas, Texas
  - Benchmark Research, Fort Worth, Texas
  - Benchmark Research, San Angelo, Texas
  - Commonwealth Clinical Research Specialist, Richmond, Virginia
  - National Clinical Research Inc., Richmond, Virginia
  - Radiant Research, Lakewood, Washington